CLINICAL TRIAL: NCT06014398
Title: Improving Survivorship and Health-related Quality of Life in Patients With Primary Brain Tumours
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Royal College of Surgeons, Ireland (Other)
Collaborators: Beaumont Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 23-127
Record Dates: First submitted 2023-07-24; First posted 2023-08-28 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-07

CONDITIONS: Hypopituitarism; Radiotherapy-Induced Hypopituitarism; Brain Tumor
MeSH Terms: conditions — Hypopituitarism; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study investigation (Experimental): All enrolled patients will undergo standardised pituitary hormone assessments.
  Interventions: Diagnostic Test: Dynamic testing of Pituitary Function

INTERVENTIONS:
Diagnostic Test: Dynamic testing of Pituitary Function — Pituitary Function Assessment:
  Baseline assessment of pituitary function by measuring ACTH, cortisol, FSH, LH, oestrogen (in females), testosterone (in males), sex hormone binding globulin, thyroid function tests, prolactin and IGF-1].
  Dynamic testing of pituitary function:
  * Patients will undergo dynamic testing of the ACTH and growth hormone axes using a glucagon stimulation test (GST).
  * Patients whose GST identifies cortisol deficiency will undergo a short synacthen test to confirm adrenal insufficiency as the GST has a false positive rate of approximately 20% for ACTH deficiency.

SUMMARY:
Background:

Approximately 480 primary, non-pituitary, brain tumours were diagnosed in Ireland each year between 1994 and 2013. Recent developments in treatment have greatly improved survival for younger patients in the 15-54 age range. The Irish National Neurosurgical Centre and the St Luke's Radiation Oncology Centre at Beaumont Hospital and treat approximately 200 patients with brain tumours per year with a combination of surgery, radiotherapy (RT) and chemotherapy with RT being the most commonly used treatment modality. With improved survivorship, the prospect of individuals living for several decades with co-morbidities induced by the tumour itself or surgical and RT treatments, raises new and complex issues for patients and clinicians.

The hypothalamus and pituitary gland in the brain are the key regulators of hormone action. They control several hormone systems including reproductive function (FSH, LH) growth (growth hormone), thyroid (TSH) and adrenal function (ACTH) as well as many other homeostatic mechanisms. It has long been recognised that therapeutic cranial RT to the pituitary gland causes hypothalamic-pituitary dysfunction (hypopituitarism). Traditionally, high-risk groups for post-irradiation hypopituitarism were considered to be patients with pituitary tumours, survivors of childhood cancer and patients who received high-dose RT to treat nasopharyngeal cancers. The potential for cranial radiotherapy to cause significant pituitary dysfunction in adult patients with brain tumours has received little attention. The assumption has been that the hypothalamic-pituitary axis is more resistant in adults than in children to the effect of cranial RT. However, it is likely that the higher doses of RT, used to treat primary brain tumours in adults, causes significant hypothalamic-pituitary dysfunction resulting in hypopituitarism. Preliminary data from the National Pituitary Centre in Beaumont Hospital has revealed that adult patients, treated with cranial radiotherapy for primary, non-pituitary brain tumours, are at risk of hypopituitarism. Approximately 40% of patients had pituitary deficiencies in at least one hormone axis, while 25% of patients had deficiencies in multiple hormone axes. Hypopituitarism confers significant morbidity and increased mortality to patients. At present, adult survivors of brain tumours are referred to the pituitary service for assessment on an ad-hoc basis meaning that many patients with hypopituitarism may go undiagnosed.

In addition to the challenges caused by hypopituitarism, long-term neuropsychological outcomes following a brain tumour cause significant functional impairments and reduced HR-QOL. Patients can present with impairments in specific cognitive domains such as memory and executive functioning or more global systems such as attention as well as significant issues with fatigue. In addition to these primary deficits, patients can also present with significant distress, fluctuant mood and anxiety. Despite the impact of brain tumours can exert, the National Cancer Control Program's National Survivorship Needs Assessment Review (2019) did not identify any studies reporting the needs of adult survivors of brain tumours in Ireland.

There is an urgent need to understand the impact of hypopituitarism and its treatment on HR-QOL and neuropsychological functioning. The proposed study will add to the limited existing literature on the prevalence of hypopituitarism in adult survivors of brain tumours treated with radiotherapy and generate detailed information on deficiency rates for individual pituitary hormones and how these deficiencies emerge over time. This will also be the first study to examine if treatment of radiotherapy-induced hypopituitarism (as part of routine clinical care) is associated with improved HR-QOL and neuropsychological functioning.

DETAILED DESCRIPTION:
Hypothesis Adult survivors of primary, non-pituitary brain tumours have an increased risk of hypopituitarism and experience impairments in HR-QOL and neuropsychological functioning. We hypothesise that diagnosis of these deficiencies and the subsequent active replacement of pituitary hormone deficits (as part of routine clinical care) will lead to an improvement in neuropsychological functioning and HR-QOL in adult survivors of primary brain tumours.

Objectives:

1. To examine the impact of radiotherapy on pituitary hormone function in adult survivors of primary, non-pituitary brain tumours.
2. To assess HR-QOL and neuropsychological functioning in adult survivors of primary, non-pituitary brain tumours.
3. To examine the impact of pituitary hormone replacement and optimisation (as part of routine clinical care) on HR-QOL and neuropsychological functioning in adult survivors of primary, non-pituitary brain tumours.

   Methods

   Study Design & Setting:

   A cross-sectional study will be conducted in the RCSI clinical research centre, located on the Beaumont Hospital campus. The study will be conducted over three years from September 2023 to September 2025.

   Participants:

   The study population will consist of adults who have previously received cranial radiotherapy for a primary, non-pituitary brain tumour.

   Patient Recruitment:
   * Participants will be identified in Professor Clare Faul's, Dr David Fitzpatrick's and Dr Nazmi ElBeltagi's clinic in St Luke's Radiation Oncology Centre at Beaumont Hospital.
   * Patients will be approached by the research fellow during routine clinical consultations.
   * The nature, purpose, benefits and risks of the study will be discussed with potential participants. They will be given the opportunity ask questions about the study. The patients' medical history will be reviewed to ensure they meet the study inclusion criteria.
   * Patients will be given a patient information leaflet and asked to read this at home.
   * The research fellow will follow up with a phone call within 72 hours and offer patients the opportunity to participate in the study. A first research study visit will be arranged for those who agree to participate.

   Study Procedure

   Study Visit One:

   Consent:
   * Participants will be asked to attend study visit one in the RCSI Clinical Research Centre (CRC).
   * Participants will be given the opportunity to ask questions and to have any concerns addressed by the research team.
   * They will then be asked by the research fellow to provide their informed consent to (i) participate in the study and (ii) allow their data to be processed by the research team.

   Assessments:
   * Participants will be asked to fast from midnight the previous evening as per Beaumont Hospital protocol for dynamic testing of pituitary function.
   * They will be advised to take their usual medications with a small sip of water on the morning of the test.
   * The research fellow will assess the participants' blood pressure, height, weight and body composition (using the bioimpedance technique with the Tanita® BC-418 segmental body composition analyser).
   * Women of childbearing age will be questioned to ensure they are not pregnancy. If there is any uncertainty, they will be asked to take a pregnancy test.

   Baseline blood sampling:
   * A fasting 9am blood sample will be taken to assess pituitary function [ACTH, cortisol, FSH, LH, oestrogen (in females), testosterone (in males), sex hormone binding globulin, thyroid function tests, prolactin, IGF-1] and metabolic phenotype [full blood count, renal/ liver profile, cholesterol, HbA1c, homeostatic model assessment for insulin resistance (HOMA-IR)].

   Dynamic testing of pituitary function:

   • Patients will undergo dynamic testing of the ACTH and growth hormone axes using a glucagon stimulation test (GST).

   • The Beaumont Hospital GST protocol will be followed throughout.

   • A cannula will be inserted into the patient's forearm. Baseline serum samples for glucose, cortisol and growth hormone will be drawn from the cannula.
   * Glucagon will then be injected into the lateral aspect of the mid quadriceps (vastus lateralis) by the research nurse/ fellow. A glucagon dose of 1mg will be used in adults less than 90kg and 1.5mg in adults greater than 90kg.
   * Serum samples will be drawn from the cannula for glucose, cortisol and GH at 90, 120, 150 and 180 minutes.

   Neuropsychological assessment:

   • A battery of neuropsychological tests to assess for cognitive, memory, language and visuo-spatial dysfunction will be performed. These tests are fully validated and have been widely used in the research setting.
   * Cognitive dysfunction: Stroop colour-word test, phonemic verbal fluency, backward digital span
   * Language dysfunction: Boston naming test
   * Memory dysfunction: Logical memory, verbal paired associate and auditory delayed recognition task
   * Visuo-spatial dysfunction Rey-osterrieth complex figure test

   HR-QOL assessment:
   * Participants' HR-QOL will be measured using extensively validated assessment tools including the Short Form-36 (SF-36), Nottingham Health Profile and EQ-5D-5L.
   * The SF-36 is a widely used HR-QOL assessment tool consisting of 4 physical and 4 mental domains which are combined to give physical and mental component summary scores. The Nottingham Health Profile consists of two components; a subjective assessment of their general health and the impact on their activities of daily living. The EQ-5D-5L assesses level of difficulty with five aspects of daily living.
   * The research fellow will ask participants the assessment questions, document their responses and calculate the overall scores (where necessary).

   Study visit one is then complete.

   Review of Pituitary Assessments:

   • Baseline and dynamic test results will be reviewed after study visit one by the principal investigator and research fellow.

   • Selected patients whose GST identifies cortisol deficiency will be asked to attend the RCSI-CRC for an additional study visit to undergo a short synacthen test (SST). This is to confirm adrenal insufficiency as the GST has a false positive rate of approximately 20% for ACTH deficiency.
   * A SST involves a cannula being inserted into the forearm and baseline serum samples for ACTH and cortisol being taken. Synacthen® 250mcg will then be administered intravenously. A second cortisol sample will be taken after 30 mins.
   * Patients diagnosed with hypopituitarism will have their hormone deficits replaced as per best clinical practice by the endocrinology service. In the event of a patient being diagnosed with growth hormone deficiency, growth hormone replacement will be discussed with the radiation oncology team is not appropriate in all types of brain tumours.
   * Patients will be counselled on the diagnosis of hypopituitarism and any questions or concerns addressed.
   * Follow up blood tests may be required to assess the adequacy of pituitary hormone replacement, as per routine clinical practice.

   Treatment History and Radiotherapy Dose Calculation:

   • The patient's tumour histology, staging and neurosurgical treatment history will be obtained from their physical and electronic medical records in Beaumont Hospital and St Luke's Centre Radiation Oncology at Beaumont Hospital.

   • The type, dose, dose per fraction of radiotherapy received by the hypothalamus/ pituitary (which will be estimated from planning scans using the biological equivalent dose) will be recorded in collaboration with Professor Clare Faul, Dr David Fitzpatrick's and Dr Nazmi ElBeltagi's in St Luke's Radiation Oncology Centre at Beaumont Hospital.

   Study Visit Two • All study participants will be asked to return for a second study visit, four months after their first visit.
   * Repeat measurements will be taken including:

     o Weight, blood pressure and body composition.

     o Fasting 9am blood samples to assess baseline pituitary function and metabolic phenotype [as previously outlined].
   * All patients will have their HR-QOL and neuropsychological functioning reassessed to measure the change over the course of the study.

   End of study

   • Patients diagnosed with hypopituitarism during the study will be followed up in the endocrinology clinic in Beaumont Hospital (as is the case for all patients with hypopituitarism).

ELIGIBILITY:
Inclusion Criteria:

* Adults (at least 18 years old) with a history of a primary, non-pituitary brain tumour which was previously treated with radiotherapy.
* Participants must have been at least 16 years old at the time of undergoing radiotherapy.
* A minimum of one year has elapsed since radiotherapy was completed.
* Capacity and willingness to provide informed consent.

Exclusion Criteria:

* Diagnosed with malignant astrocytic brain tumour with life expectancy of less than six months.
* Brain tumour infiltration of the hypothalamus or pituitary pre-operatively.
* Previously diagnosis of hypopituitarism.
* Oral glucocorticoid use within the last three months.
* Pregnant or breastfeeding women at the time of recruitment.
* Unable to provide informed consent for inclusion in this study.
* Opinion of the radiation oncology or research team that participation in the study is not in the best interest of the patient for any reason.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of radiotherapy-induced hypopituitarism | Assessed at Baseline
  Prevalence of pituitary hormone deficiencies in adult survivors of primary, non-pituitary brain tumours, previously treated with radiotherapy.

SECONDARY OUTCOMES:
HR-QOL | Assessed at baseline
  The Short Form-36 will be used to assess HR-QOL in the study population relative to a published normative population. The SF-36 is a generic questionnaire consisting of 8 domains; physical function, bodily pain, role physical, general health, vitality, social functioning, role emotional, mental health. Each domain is scored form 0-100, with higher scores indicating better quality of life.
Change in HR-QOL | Assessed at 4 months
  HR-QOL will be reassessed at 16 weeks using the SF-36 in (i) participants with hypopituitarism and (ii) participants with normal pituitary function. The SF-36 is a generic questionnaire consisting of 8 domains; physical function, bodily pain, role physical, general health, vitality, social functioning, role emotional, mental health. Each domain is scored form 0-100, with higher scores indicating better quality of life.

CONTACTS AND LOCATIONS:
Locations (2):
- Ireland (2):
  - Beaumont Hospital, Dublin
  - St Luke's Radiation oncology Centre, Beaumont Hopsital, Dublin

IPD SHARING:
Plan to Share IPD: No